CLINICAL TRIAL: NCT05916885
Title: Effects of Short-intensity Modified Constraint-induced Movement Therapy on Hand Function in Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0213
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Hemorrhagic Stroke; Ischemic Stroke; Rehabilitation
Keywords: Hemorrhagic Stroke; Ischemic Stroke; Rehabilitation
MeSH Terms: conditions — Hemorrhagic Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be allocated into two groups by randomization. The experimental group in which patients will be given short-intensity mCIMT along with conventional therapy. A control group, in which patients will be given conventional therapy alone. The therapy regime will be 3 hours/ day, 5 days/week, and 4 successive weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): an experimental group receiving short-intensity modified CIMT and conventional therapy
  Interventions: Other: short-intensity modified CIMT and conventional therapy
- control group (Active Comparator): a control group receiving conventional therapy alone.
  Interventions: Other: conventional therapy alone

INTERVENTIONS:
Other: short-intensity modified CIMT and conventional therapy — an experimental group receiving short-intensity modified CIMT and conventional therapy
  Arms: experimental group
Other: conventional therapy alone — a control group receiving conventional therapy alone.
  Arms: control group

SUMMARY:
To determine effects of short-intensity modified constraint-induced movement therapy on hand function in stroke patients.

DETAILED DESCRIPTION:
The aim of the study is to determine the effects of a short-intensity modified CIMT (mCIMT) program on hand function in stroke patients. This study will be a randomized controlled trial comprising two groups, an experimental group in which patients will be given short-intensity mCIMT along with conventional therapy. A control group, in which participants will be given conventional therapy alone. Patients will be assessed with the Wolf Motor Function Test, the Motor Activity Log, and the Ashworth Scale before and after treatment. The data will be analyzed by using SPSS for windows software version 25. Statistical significance will be set at p=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients having the First stroke either ischemic or hemorrhagic (3-24 months after stroke)
* Patients having Mini-mental status examination score (MMSE) ≤23/30
* Patients having Passive range of motion (PROM) includes at least 90 degrees shoulder flexion and abduction, 45degrees shoulder external rotation,- 30 degrees elbow extension, and 45 degrees forearm supination and pronation (from a neutral position). At least 10 degrees active wrist extension, 10 degrees abduction/thumb extension, and 10-degree extension at the level of the metacarpophalangeal and interphalangeal joints between the two toes among the II-III-IV-V fingers (these movements will be repeated starting from a resting position 3 times in 1 minute).

Exclusion Criteria:

* Patients having Subarachnoid hemorrhage.
* Patients having Motor activity log - the amount of use score ≥2.5
* Patients having treatment of upper limb spasticity (e.g., botulinum toxin) in the 3 months prior to the start of the study and/or during its execution.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Wolf motor function test (WMF) | 9 months
  Wolf motor function test (WMF) is a new time-based method for evaluating upper extremity performance that provides insight into joint-specific and whole limb movements.
  To investigates the effects of mandatory exercise therapy in patients with mild to moderate stroke and traumatic brain injury. The original version of the WMFT consisted of 21 items.
  The widely used WMFT consists of 17 items. The first 6 items consist of timed functional tasks, items 7 and 14 measure muscle strength, and the remaining 9 items consist of analyses of the quality of movement in accomplishing various tasks.
The motor activity log | 9 months
  The motor activity log is a structured interview, designed to explore how and how well subjects are using the more affected arm outside of a laboratory setting. Participants are asked standardized questions about their high-impact arm usage (amount scale or AS) and quality of movement (how good scale or HW) during a specified functional activity. The scale is printed on a separate sheet and placed in front of the participant during test administration.
  Participants should be told that they can give half marks (i.e. 0.5, 1.5, 2.5, 3.5, 4.5) if this reflects their assessment.
The Ashworth scale, | 9 months
  The Ashworth scale, which rates each passive movement between 1 (normal) and 5 (immobility), was used in a recent study and is easier to use than other methods and applicable to wide-range movements.

CONTACTS AND LOCATIONS:
Overall Officials: Zeest Hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tedla JS, Gular K, Reddy RS, de Sa Ferreira A, Rodrigues EC, Kakaraparthi VN, Gyer G, Sangadala DR, Qasheesh M, Kovela RK, Nambi G. Effectiveness of Constraint-Induced Movement Therapy (CIMT) on Balance and Functional Mobility in the Stroke Population: A Systematic Review and Meta-Analysis. Healthcare (Basel). 2022 Mar 8;10(3):495. doi: 10.3390/healthcare10030495. PMID 35326973
- [Background] Uswatte G, Taub E, Lum P, Brennan D, Barman J, Bowman MH, Taylor A, McKay S, Sloman SB, Morris DM, Mark VW. Tele-rehabilitation of upper-extremity hemiparesis after stroke: Proof-of-concept randomized controlled trial of in-home Constraint-Induced Movement therapy. Restor Neurol Neurosci. 2021;39(4):303-318. doi: 10.3233/RNN-201100. PMID 34459426
- [Background] Takebayashi T, Takahashi K, Moriwaki M, Sakamoto T, Domen K. Improvement of Upper Extremity Deficit after Constraint-Induced Movement Therapy Combined with and without Preconditioning Stimulation Using Dual-hemisphere Transcranial Direct Current Stimulation and Peripheral Neuromuscular Stimulation in Chronic Stroke Patients: A Pilot Randomized Controlled Trial. Front Neurol. 2017 Oct 30;8:568. doi: 10.3389/fneur.2017.00568. eCollection 2017. PMID 29163334